CLINICAL TRIAL: NCT03623230
Title: Concentration-Volume Relationship of Bupivacaine in Femoral Nerve Block Efficiency for Postoperative Analgesia in Primary Total Knee Arthroplasty: A Randomized Controlled Double Blind Clinical Trial
Brief Title: Concentration Effect of Local Anesthetics on Femoral Nerve Block Efficiency
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bozyaka Training and Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DizFemoralKonsant
Record Dates: First submitted 2018-06-30; First posted 2018-08-09 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Anesthesia, Conduction; Arthroplasty, Replacement, Knee; Pain, Postoperative; Anesthesia and Analgesia
Keywords: Femoral nerve block; peripheral nerve block; Concentration; volume; bupivacaine; post operative analgesia; total knee arthroplasty
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Anesthesia, Conduction; Bandages; Bupivacaine

STUDY DESIGN:
Intervention Model Description: Three groups involved. One control group and two nerve block groups with different drug concentration
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- GCont (Sham Comparator): Only dressing will be applied to patients without actually nerve block performed
  Interventions: Other: Dressing
- G125 Block (Active Comparator): Ultrasound Guided Femoral Nerve Block: 20ml Bupivacaine 0.125% Injectable Solution will be administered for femoral nerve block.
  5ml %0,5 Bupivacaine will be diluted with 15ml Saline solution.
  Interventions: Procedure: Ultrasound Guided Femoral Nerve Block; Drug: Bupivacaine 0.125% Injectable Solution
- G25 Block (Active Comparator): Ultrasound Guided Femoral Nerve Block: 10ml Bupivacaine 0.25% Injectable Solution will be administered for femoral nerve block.
  5ml %0,5 Bupivacaine will be diluted with 5ml Saline solution.
  Interventions: Procedure: Ultrasound Guided Femoral Nerve Block; Drug: Bupivacaine 0.25% Injectable Solution

INTERVENTIONS:
Procedure: Ultrasound Guided Femoral Nerve Block — Femoral nerve block will be applied post-operatively with guidance of USG and nerve stimulator
  Other Names: Regional Anesthesia
  Arms: G125 Block; G25 Block
Other: Dressing — Only dressing will be applied to related area to protect blindness between groups
  Arms: GCont
Drug: Bupivacaine 0.25% Injectable Solution — Perineural Injection
  Other Names: Marcaine
  Arms: G25 Block
Drug: Bupivacaine 0.125% Injectable Solution — Perineural Injection
  Other Names: Marcain
  Arms: G125 Block

SUMMARY:
US-guided femoral nerve block is used effectively in post-operative pain management in the surgical treatment of the lower extremity. However, the volume and concentration of the local anesthetic drug to be administered remains controversial. In this prospective, randomized, double-blinded study, patients who underwent unilateral primary total knee arthroplasty and successfully performed spinal anesthesia with standard method and dosage, will be selected for US-guided femoral nerve block after the operation. Patients will be divided into three groups with simple randomization. The First group will be determined as the control group (GCont) and only dressing will be applied to the patients. For second group(G125), 0,125% 20 ml local anesthetic and for the third group (G25), 0,25% 10 ml local anesthetic will be administered to the femoral nerve without changing the drug dose (25 mg bupivacaine). Whether there is a difference between post-op analgesia durations, motor block formation, mobilization time and 90° flexion time between the groups will be investigated.

DETAILED DESCRIPTION:
All patients scheduled for total knee arthroplasty will be evaluated before the operation. Eligible patients will be informed about the study and "Numeric Rating Scale" for pain evaluation. Then, patients will be asked for informed consent. After approval from the local research ethics committee, first patient will be recruited for study and patient's group will be determined by dice roll(1,4: GCont - 2,5: G125 - 3,6: G25). Patients who are scheduled for primary total knee arthroplasty under spinal anesthesia with a planned sensory block level between T4 and T7 dermatomes, will be recruited and assigned to a group. After successfully completed surgery, patients will be administered femoral nerve block or only dressing according to the relevant group. Before femoral nerve block is performed, patients will be re-informed about Numeric Rating Scale(NRS) and will be asked to rate their pain at the moment.

* Control Group(GCont) patients will only be applied sterile dressing for the purpose of blinding the patient and the follow-up physician.
* 0.125% Bupivacaine Group(G125) patients will be administered femoral block with 20 ml 0.125% Bupivacaine by an experienced anesthesiologist.
* 0.25% Bupivacaine Group(G25) patients 10ml will be administered femoral block with 0.25% Bupivacaine by an experienced anesthesiologist.

The procedures will be performed in the operating room under both US and nerve stimulator guidance. Patients will be followed-up in post-anesthesia care unit and in the ward for 48 hours. Scheduled and on-demand(Tramadol) medication for analgesia will be ordered and nurses will be informed about the study. Patients' pain scores and ambulation times will be followed-up by another anesthesiologist and on-demand medication will be recorded and monitored from hospital's computer based hospital management program online. Patients will be followed-up for six months after the surgery in order to explore potential long term benefits and complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are scheduled for primary unilateral total knee arthroplasty under spinal anesthesia
* Patients who has informed consent for study

Exclusion Criteria:

* Patient's refusal to participate
* Patients under 18 years of age
* Patients who are undergoing surgery with an anesthesia technique other than spinal anesthesia for any reason (general anesthesia, laryngeal mask application, etc.)
* Patients with known local anesthetic allergy
* Patients with Body mass index > 35
* Patients diagnosed sepsis and bacteriemia,
* Skin infection at the injection site,
* History of coagulopathy or anticoagulant therapy
* Patients with uncontrolled diabetes ,
* Uncoordinated patients,
* Psychological and emotional lability,
* Surgical intervention longer than 3 hours.
* Patients with pre-operative limitation of movement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2018-08-10 (Actual); Primary Completion 2018-12-12 (Actual); Study Completion 2019-02-15 (Actual)

PRIMARY OUTCOMES:
Post-operative pain assessed by Numeric Rating Scale (NRS) | 30th minute postoperatively
  Pain scores will be recorded as reported by the patient according to NRS
Post-operative pain assessed by Numeric Rating Scale (NRS) | 1st hour postoperatively
  Pain scores will be recorded as reported by the patient according to NRS
Post-operative pain assessed by Numeric Rating Scale (NRS) | 2nd hour postoperatively
  Pain scores will be recorded as reported by the patient according to NRS
Post-operative pain assessed by Numeric Rating Scale (NRS) | 6th hour postoperatively
  Pain scores will be recorded as reported by the patient according to NRS
Post-operative pain assessed by Numeric Rating Scale (NRS) | 12th hour postoperatively
  Pain scores will be recorded as reported by the patient according to NRS
Post-operative pain assessed by Numeric Rating Scale (NRS) | 24th hour postoperatively
  Pain scores will be recorded as reported by the patient according to NRS
Post-operative pain assessed by Numeric Rating Scale (NRS) | 48th hour postoperatively
  Pain scores will be recorded as reported by the patient according to NRS

SECONDARY OUTCOMES:
Ambulation Time | 72 hours post-operatively
  First time a patients can walk around independently
Opioid Consumption | 48 hour post-operatively
  Opioids(Tramadol) will be administered to patients in case demanded.

OTHER OUTCOMES:
Long Term Infection | Six months post-operatively
  Surgery site or prosthesis infection in six months following surgery

CONTACTS AND LOCATIONS:
Overall Officials: Zeki T TEKGUL, Associate Professor, Study Director — Izmir Bozyaka Training and Research Hospital
Locations (1):
- Izmir Bozyaka Training and Research Hospital, Karabağlar, İzmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Karlsen AP, Wetterslev M, Hansen SE, Hansen MS, Mathiesen O, Dahl JB. Postoperative pain treatment after total knee arthroplasty: A systematic review. PLoS One. 2017 Mar 8;12(3):e0173107. doi: 10.1371/journal.pone.0173107. eCollection 2017. PMID 28273133
- [Background] Tulgar S, Selvi O, Senturk O, Serifsoy TE, Sanel S, Meydaneri S. Evaluation of analgesic regimens in total knee arthroplasty, retrospective study. North Clin Istanb. 2017 Aug 25;4(2):124-130. doi: 10.14744/nci.2017.88598. eCollection 2017. PMID 28971169
- [Background] Thobhani S, Scalercio L, Elliott CE, Nossaman BD, Thomas LC, Yuratich D, Bland K, Osteen K, Patterson ME. Novel Regional Techniques for Total Knee Arthroplasty Promote Reduced Hospital Length of Stay: An Analysis of 106 Patients. Ochsner J. 2017 Fall;17(3):233-238. PMID 29026354